CLINICAL TRIAL: NCT00105352
Title: Improving Metabolic Assessments in Type 1 Diabetes Mellitus Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Juvenile Diabetes Research Foundation (Other); National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MMTTGST (IND) (completed)
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes Study Group; TrialNet; type 1 diabetes; juvenile onset diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Procedure: Mixed Meal Tolerance Test
Procedure: Glucagon Stimulation Test

SUMMARY:
OBJECTIVE:

This study is being conducted by the Type 1 Diabetes TrialNet Study Group, funded by the National Institutes of Health, in collaboration with the European C-Peptide Group. The goal is to evaluate comparability and reproducibility of measures of beta cell function in type 1 diabetes comparing the mixed meal tolerance tests (MMTT) and glucagon stimulation test (GST). These two tests will be compared to assess the relationship between the MMTT and IV (intravenous) Glucagon stimulated C-peptide responses as measured by time to peak C-peptide and AUC (area under the curve) values.

Based on the understanding that type 1 diabetes results from an immune mediated loss of pancreatic beta cells, therapeutic trials and newer measures of beta cell function can be evaluated as endpoints for clinical trials. Direct assessment of residual beta cell function is an appropriate endpoint, as retention of beta cell function in patients with T1D is known to result in improved glycemic control and reduced hypoglycemia, retinopathy and nephropathy. Endogenous beta cell function or insulin secretion is best measured by determination of C-peptide (which is co-secreted with insulin in a 1:1 molar ratio). Intervention studies over the past few decades have usually used measurement of C-peptide. However, the relationship between these or other measures of beta cell function has not been well studied. The relative advantages of one measure over another in terms of variability, sensitivity and burden to the subject is unknown. In addition, the optimal conditions for the conduct of the test need to be determined.

An important goal is to develop an international consensus about the conduct of metabolic tests in the context of large, multicenter trials involving type 1 diabetes (T1D) by balancing the scientific data with the burden on the subject.

DETAILED DESCRIPTION:
Overview:

The study is a multi-center, two-arm, randomized clinical trial. Each participant will undergo four tests within a limited period according to the test sequence assignment. The tests will randomly start with either MMTT or GST.

Specific Aims

* To compare the reliability of the MMTT and Glucagon stimulated C-peptide responses as measured by time to peak C-peptide on MMTT, and the peak and AUC values on both tests.
* To determine the relationship between MMTT and Glucagon stimulated C-peptide responses as measured by time to peak C-peptide on MMTT and peak and AUC values on both tests.
* To determine the impact of basal glucose, peak glucose, age of participant, time from diagnosis, and basal C-peptide with respect to the reliability of measures and relationship between MMTT and Glucagon results.
* Describe the palatability of, patient compliance with, and adverse effects of each test (MMTT vs. GST) and to compare the participant and investigator burden to conduct the MMTT and Glucagon tests.

TEST INFORMATION:

* Mixed Meal Tolerance Test (MMTT):

BOOST is a liquid meal (like a milkshake) containing a standard amount of fat, protein, and carbohydrate. BOOST raises blood sugar and causes the pancreas to produce insulin. After drinking BOOST, about one-half teaspoon of blood will be drawn through an IV line in the arm after 15, 30, 60, 90, and 120 minutes. (Using an IV line avoids multiple needle sticks). The test takes about 2 hours.

* Glucagon Stimulation Test (GST):

Glucagon is a hormone that circulates in the blood and stimulates insulin secretion. Glucagon will be injected into the bloodstream through an IV line, and about one-half teaspoon of blood will be drawn five times during ten minutes. The test takes about 30 minutes.

OTHER TEST INFORMATION:

* Participants will have tests on four different days over a six week period. Participants will have either a) two MMTTs and then two GSTs OR b) two GSTs and then two MMTTs. Each test will be done 3-10 days apart.
* Participants will follow a special high carbohydrate diet (150 grams) for at least three days prior to each study visit. Dietary information will be provided.
* Participants will fast overnight (at least 8 hours) and arrive at the clinic between 7 AM - 10 AM.
* It is essential that participants have a blood glucose level of 70-200 mg/dl in the morning before starting the test. If blood glucose is too high or too low the morning of the test, the test will be re-scheduled on another day.
* Tests will be re-scheduled if, on the morning of the test, your blood sugar or ketones are not within acceptable ranges. Testing could take up to eight visits if tests need to be re-scheduled.
* Participants will learn whether their pancreas is still secreting insulin and, if so, how much insulin is being secreted. This information may help their diabetes health care team design for them a better insulin regimen and diabetes management program to improve their longterm blood sugar control.
* This study will help researchers learn which test (MMTT or GST) is best to use in other research studies looking at treatments that may stop or delay type 1 diabetes.

ELIGIBILITY:
* Informed consent obtained from participants (over 12 years of age) and parents (for participants below 18 years of age). Assent is obtained from younger children.
* Age 8 - 35 years at the time of inclusion
* Body weight > 30 kg
* Type 1 diabetes defined by: ADA (American Diabetes Association) criteria or judgment of physician
* Duration of diabetes: 1 month to 3* years (*The TrialNet Coordinating Center will monitor fasting C-peptide levels as they are reported to ensure that a wide range of values is included. This review may result in widening the duration of diabetes window to allow for subjects with low C-peptide).
* Must maintain good glycemic control
* Be willing to travel to a TrialNet Clinical Center for a minimum of four separate visits that are spaced 3-10 days apart, and be willing to complete the study within a six week period.

Exclusion Criteria:

* Actual treatment with drugs influencing beta cell function (e.g. oral hypoglycaemic agents, beta-2-receptor agonists)
* Actual treatment with drugs influencing insulin sensitivity (e.g. steroids)
* Significant concomitant disease likely to interfere with glucose metabolism (e.g. febrile illness within the prior 3 days)
* Expected poor compliance
* If a female of child-bearing age, currently pregnant or not using a form of birth control
* Any other condition that by the judgement of the investigator may be potentially harmful to the patients

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2004-11; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Stimulated C-peptide response derived from the 2-hour MMTT and the glucagon stimulation test (GST)
Time to peak C-peptide on MMTT, and the peak and AUC values from each test
Co-efficient of reproducibility of the MMTT, and the GST, provided from the duplicate tests within the same individuals

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Skyler, M.D., Study Chair — University of Miami
Locations (18):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Riley Hospital for Children, Indiana University, Indianapolis, Indiana
  - Joslin Diabetes Center/ Children's Hospital Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Naomi Berrie Diabetes Center, Columbia University, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Medical Center at Dallas, Dallas, Texas
  - Benaroya Research Institute, Seattle, Washington
- Walter and Eliza Hall Institute of Medical Research, Parkville, Victoria, Australia
- University of Toronto, Toronto, Ontario, Canada
- University of Turku, Turku, Finland
- Vita-Salute San Raffaele University, Milan, Italy
- University of Bristol, Bristol, United Kingdom

REFERENCES:
- [Background] Palmer JP, Fleming GA, Greenbaum CJ, Herold KC, Jansa LD, Kolb H, Lachin JM, Polonsky KS, Pozzilli P, Skyler JS, Steffes MW. C-peptide is the appropriate outcome measure for type 1 diabetes clinical trials to preserve beta-cell function: report of an ADA workshop, 21-22 October 2001. Diabetes. 2004 Jan;53(1):250-64. doi: 10.2337/diabetes.53.1.250. PMID 14693724
- [Background] Greenbaum CJ, Harrison LC; Immunology of Diabetes Society. Guidelines for intervention trials in subjects with newly diagnosed type 1 diabetes. Diabetes. 2003 May;52(5):1059-65. doi: 10.2337/diabetes.52.5.1059. No abstract available. PMID 12716733
- [Derived] Greenbaum CJ, Mandrup-Poulsen T, McGee PF, Battelino T, Haastert B, Ludvigsson J, Pozzilli P, Lachin JM, Kolb H; Type 1 Diabetes Trial Net Research Group; European C-Peptide Trial Study Group. Mixed-meal tolerance test versus glucagon stimulation test for the assessment of beta-cell function in therapeutic trials in type 1 diabetes. Diabetes Care. 2008 Oct;31(10):1966-71. doi: 10.2337/dc07-2451. Epub 2008 Jul 15. PMID 18628574
- See also: TrialNet Study Group — http://diabetestrialnet.org
- See also: American Diabetes Association — http://www.diabetes.org
- See also: Juvenile Diabetes Research Foundation, International — http://jdrf.org